CLINICAL TRIAL: NCT00322777
Title: A Spirituality Teaching Program for Depression in Adults: A Randomized Controlled Trial
Brief Title: Spirituality Teaching Program for Depressed Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Institute of Natural and Integrative Medicine (Other)
Collaborators: University of Calgary, Dept. of Psychiatry & Dept. of Community Health Sciences (Unknown); Southwest Behavioral Health Sciences (Unknown); Alberta Health services (Other); Arizona School of Health Sciences (Other); The Center for Mind-Body Medicine (Other)
Responsible Party: Principal Investigator, Badri Rickhi, Chair and Founding Member, CINIM, Canadian Institute of Natural and Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Spirit II
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Major Depression
Keywords: Major depression; Spirituality; Randomized clinical trial
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirituality Group (Experimental): Arm where participants began the intervention (the Spirituality Teaching Program) upon recruitment for an 8 week period. Therefore, the program was initiated at week 1 of the trial.
  Interventions: Behavioral: Spirituality Teaching Program
- Waitlist Control Group (Active Comparator): Arm where participants began the intervention (the Spirituality Teaching Program) after an 8 week wait period. Therefore, the program was initiated at week 8 of the trial. Between week 1 and week 8, participants did not complete the program and were instructed to carry out their day to day activities as before.
  Interventions: Behavioral: Spirituality Teaching Program

INTERVENTIONS:
Behavioral: Spirituality Teaching Program — The Spirituality Teaching Program is a home study program delivered through audio CDs over an 8-week period. The program consists of weekly 90 minute teaching sessions, based on the content of a workshop developed to assist users in developing a more spiritual outlook on life and coping resources. Using didactic comment and storytelling, the following spiritual concepts are addressed in the sessions: self-transcendence, connectedness, forgiveness, self-acceptance, detachment, compassion and gratitude. Each session concludes with a relevant guided visualization practice. In addition, a 15-minute progressive relaxation exercise is included that is to be used on a daily basis. The presented content is nondenominational to ensure compatibility with any beliefs participants may hold.

SUMMARY:
Major depression is a widely spread health problem in Canada. Recent research suggests a potential role for religion/spirituality in the prevention of and recovery from depression in adults. The purpose this study was to assess the efficacy of a home-based Spirituality Teaching Program for adults in the treatment of major depression. The objectives of the study were to determine:

1. whether the Spirituality Teaching Program is efficacious in improving depression severity, response rate, and remission rate in adults,
2. whether efficacy is maintained long term (over a 16 week period).

DETAILED DESCRIPTION:
Major depression is a widely spread health problem in Canada with a life time prevalence of 11% in men and 16% in women. A recent avenue of research suggests a role for religion/spirituality in the prevention of and recovery from depression. It has been hypothesized that religion/spirituality acts as a coping resource in distressing life situations including illness and loss and may address the struggles of depressed patients of feeling separated from their surrounding world, as well as from their inner self. Majority of the research conducted to date on this topic has been observational and focused on the religious denomination, primarily the Christian and Muslim faiths. However, given the distinction between spirituality and religion and since a growing portion of the Canadian population identifies themselves as nonreligious but spiritual (10), it is pertinent to explore whether there is a role for a nondenominational spiritual intervention as a mental health resource. Considering the burden of depression on an individual and social level and need for effective and accessible treatment options, evaluation of spirituality based approaches is highly relevant. This study aims to assess whether nurturing spiritual coping resources in a non-faith based way may play a therapeutic role in recovery from major depression in adults.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy the DSM-IV criteria for unipolar major depression with a depression score of 18-22 on the Hamilton Depression Scale (mild to moderate severity),
* Are at least 18 years of age,
* Have the competence to understand the study requirements and the ability to comply with the study intervention,
* Have provided written informed consent.

Exclusion Criteria:

* History of treatment resistance to two or more antidepressants when treated for an adequate period with a therapeutic dose
* History of bipolar d/o, psychotic d/o, any psychotic episodes, personality d/o (except obsessive compulsive d/o)
* History of multiple suicide attempts
* Acute psychiatric condition other than unipolar depression
* Regular use of medications (other than antidepressant, if applicable) that have mood altering effects, such as narcotics, anticonvulsants, illicit drugs or sleeping pills
* Uncontrolled medical conditions in the last 3 months
* DSM-IV diagnosis of substance abuse (except nicotine and caffeine) within the past 12-months
* High suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Badri Rickhi, MD, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; John Toews, MD, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; Sabine Moritz, MSc, Study Director — Alberta Health Services (current)
Locations (1):
- Canadian Institute of Natural and Integrative Medicine, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moritz S, Kelly MT, Xu TJ, Toews J, Rickhi B. A spirituality teaching program for depression: qualitative findings on cognitive and emotional change. Complement Ther Med. 2011 Aug;19(4):201-7. doi: 10.1016/j.ctim.2011.05.006. Epub 2011 Jun 29. PMID 21827934
- [Result] Rickhi B, Moritz S, Reesal R, Xu TJ, Paccagnan P, Urbanska B, Liu MF, Ewing H, Toews J, Gordon J, Quan H. A spirituality teaching program for depression: a randomized controlled trial. Int J Psychiatry Med. 2011;42(3):315-29. doi: 10.2190/PM.42.3.f. PMID 22439299

RESULTS

PARTICIPANT FLOW:
Groups:
- Waitlist Control Group: Arm where participants began the intervention (the Spirituality Teaching Program) after an 8 week wait period. Therefore, the program was initiated at week 8 of the trial. Between week 1 and week 8, participants were instructed to carry out their day to day activities as before.
Period: Overall Study
Arm/Group | Spirituality Group | Waitlist Control Group
Started | 39 | 45
Data Collection at BASELINE| | 39 | 45
Data Collection at Week 8 | 39 | 45
Data Collection at Week 16 | 39 | 45
Data Collection at Week 24 | 39 | 45
Completed | 39 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spirituality Group | Waitlist Control Group | Total
Number analyzed (Participants) | 39 | 45 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (10.86) | 44.0 (9.14) | 44.02 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 65
  Male | 10 | 9 | 19
Marital Status [Number; unit: participants]
  Married/common law | 27 | 22 | 49
  Not married | 12 | 23 | 35
Education [Number; unit: participants]
  less than or equal to Highschool | 5 | 7 | 12
  Some college or university | 9 | 8 | 17
  graduated from college or university | 22 | 24 | 46
  Postgraduate or professional degree | 2 | 6 | 8
  Not available | 1 | 0 | 1
Employment status [Number; unit: participants]
  Paid work | 31 | 33 | 64
  No paid work | 8 | 12 | 20
Religious denomination [Number; unit: participants]
  No religion | 14 | 16 | 30
  Christian | 22 | 25 | 47
  Other | 3 | 4 | 7
Interest in spirituality [Number; unit: participants]
  A little interested | 4 | 3 | 7
  Quite interested | 11 | 12 | 23
  Very interested | 24 | 30 | 54

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale - Depression Severity
Description: Depression severity was assessed at the four time points (baseline, 8 weeks, 16 weeks and 24 weeks) using the Hamilton Depression Rating Scale (HAM-D). The HAM-D is a standardized outcome measure of depression severity in adults. Total scores includes the sum of 17-items, with eight items scored on a range of 0 (absent) to 2 (marked or definite) and nine scored on a range of 0 (absent) to 4 (very severe). The level of depression was based on the following scoring ranges: 7 or under not depressed, 8-13 some depressive symptoms but no depressive disorder, 12-15 mild depression, 16-19 moderate depression, 20-24 moderately severe depression, and 25+ severe depression.
  The HAM-D was administered through a face to face interview, which was conducted by a trained nurse who was blinded to participants' allocation.
Time Frame: baseline, 8 weeks, 16 weeks, and 24 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Spirituality Group | Waitlist Control Group
Number analyzed (Participants) | 39 | 45
units on a scale
  Baseline | 20.4 [19.9 to 20.9] | 20.3 [19.8 to 20.8]
  8 weeks | 11.9 [10.2 to 13.5] | 18.0 [16.4 to 19.7]
  16 weeks | 10.7 [8.5 to 13.0] | 12.0 [9.8 to 14.2]
  24 weeks | 10.4 [8.0 to 12.7] | 10.1 [7.8 to 12.4]

2. Secondary Outcome: Response Rate
Description: Response rate was assessed at the four time points (baseline, 8 weeks, 16 weeks and 24 weeks) using the Hamilton Depression Rating Scale (HAM-D). A response was determined as a reduction in the HAM-D score by at least 50% from the baseline score. The data are presented as the percentage of participants with response at each time point as compared to baseline.
Time Frame: baseline, 8 weeks, 16 weeks, and 24 weeks
Measure: Number; unit: percentage of participants with response
Arm/Group | Spirituality Group | Waitlist Control Group
Number analyzed (Participants) | 39 | 45
percentage of participants with response
  8 weeks | 35.9 | 4.4
  16 weeks | 56.4 | 51.1
  24 weeks | 64.1 | 66.7

3. Secondary Outcome: Remission
Description: Remission of depression was assessed at the four time points (baseline, 8 weeks, 16 weeks and 24 weeks) using the Hamilton Depression Rating Scale (HAM-D). Remission was based on a HAM-D score of less than 7. Remission is indicated as a percentage of participants at each time point whose scores were below 7.
Time Frame: baseline, 8 weeks, 16 weeks, and 24 weeks
Measure: Number; unit: percentage of participants score < 7
Arm/Group | Spirituality Group | Waitlist Control Group
Number analyzed (Participants) | 39 | 45
percentage of participants score < 7
  8 weeks | 30.7 | 2.2
  16 weeks | 38.5 | 31.1
  24 weeks | 41 | 53.3

ADVERSE EVENTS:
Arm/Group | Spirituality Group | Waitlist Control Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/45
Other Adverse Events (participants affected / at risk) | 0/39 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No